CLINICAL TRIAL: NCT06221358
Title: Pharmacogenomics of Stimulant Treatment Response in Children and Adolescents With Attention-Deficit/ Hyperactivity Disorder
Brief Title: Pharmacogenomics of Stimulant Treatment Response
Acronym: PGx-STaR
Status: Recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Chad Bousman, Associate Professor, University of Calgary
Other Study IDs: REB23-0366
Record Dates: First submitted 2024-01-02; First posted 2024-01-24 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Attention-Deficit/ Hyperactivity Disorder (ADHD)
Keywords: Children; Adolescents; ADHD; Pharmacogenetics; Neurology; Psychostimulants; Methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will donate a 2 mL (teaspoon) sample of saliva and 0.07 mL (1/64th of a teaspoon) of blood via a needle-free collection device.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The "Pharmacogenomics of Stimulant Treatment Response" (PGx-STaR) study aims to identify genetic profiles related to methylphenidate treatment outcomes in children and adolescents aged 6-24 with Attention deficit/hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
Background: ADHD is a common neurodevelopmental disorder affecting children and adolescents, with psychostimulants, specifically slow-release methylphenidate (e.g., Biphentin®, Concerta®), being a first-line treatment option. However, the response to medications varies significantly among individuals, with some experiencing limited benefits or intolerable side effects. Unlike other areas of psychiatry, ADHD pharmacotherapy lacks genetic markers to guide treatment decisions, resulting in delayed symptom relief and diminished quality of life for patients.

Objectives:

1. Identifying genomic profiles associated with psychostimulant treatment response and tolerability in children and adolescents with ADHD.
2. Establishing a research platform for the discovery of new genetic and non-genetic markers of drug treatment outcomes relevant to mental health care in children.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for participation if all the following are true.

* Aged 6 - 24 years.
* Located in Western Canada (i.e., Alberta, British Columbia, Saskatchewan, Manitoba).
* Primary diagnosis of ADHD (all types).
* Starting Methylphenidate (excluding immediate release forms) treatment.

Exclusion Criteria:

Patients will be excluded from participation if any of the following are true.

* Co-occurring psychotic, bipolar or eating disorders.
* Significant risk of suicide.
* An intellectual disability, or diagnosis of autism spectrum disorder (ASD) or tics/Tourette disorders.
* Past 12-month high-risk alcohol or substance use defined as monthly or more frequent use.
* Psychotherapy or brain stimulation-based therapy initiated within 8 weeks of referral or plans to initiate/change these types of therapies during the study
* History of liver or bone marrow (hematopoietic cell) transplant as these events can result in ambiguous genomic results.

Ages: 6 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescent with primary diagnosis of ADHD (all types), aged 6-24 years.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in ADHD symptom severity | Baseline and 1, 2, 3, and 4 weeks post-baseline
  Strengths and Weaknesses of Attention-Deficit/Hyperactivity Symptoms and Normal Behavior Scale (SWAN) Rating Scale for ADHD. Score range = -90 to +90, with higher scores indicative of worse outcome.
Side effect frequency and severity | 1, 2, 3, and 4 weeks post-baseline
  CADDRA ADHD Medication and Side Effect Form

SECONDARY OUTCOMES:
Methylphenidate/ritalinic acid exposure | 4 weeks post-baseline
  Methylphenidate and ritalinic acid trough plasma levels
Change in working memory | Baseline and 4 weeks post-baseline
  Sorting Working Memory Test (7 minutes; administered orally and online with research team member). An assessment of working memory. A participant is asked to recall and sequence different stimuli that are presented visually and via audio. Higher scores indicate better outcome.
Change in attention | Baseline and 4 weeks post-baseline
  Dimension Change Card Sort Test (8 minutes; administered online). An assessment of cognitive flexibility and attention. A participant is asked to match a series of picture pairs to a target picture. Higher scores indicate better outcome.
Change in inhibitory control | Baseline and 4 weeks post-baseline
  Flanker Inhibitory Control and Attention Test (7 minutes; administered online). An assessment of inhibitory control and attention. A participant is asked to focus on a particular stimulus while inhibiting attention to the stimuli flanking it. Higher scores indicate better outcome.
Change in impulse control | Baseline and 4 weeks post-baseline
  Stop Signal Task (10 minutes; administered online). An assessment of impulse control. A participant is presented with a target stimulus and are asked to respond to the stimulus as fast as possible. Higher score indicate better outcome.
Change in functioning | Baseline and 4 weeks post-baseline
  Columbia Impairment Scale. Score range 0-52, with higher scores indicative of worse outcome.
Change in child quality of life | Baseline and 4 weeks post-baseline
  Pediatric Quality of Life Inventory (PedsQoL). Items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better quality of life.
Change in carer quality of life | Baseline and 4 weeks post-baseline
  Care-related Quality of Life instrument (Carer QoL-7D). Utility tariffs for the CarerQol have been developed to calculate a CarerQol-7D utility score from the responses on the seven dimensions, ranging between 0 ('worst imaginable caregiving situation') and 100 ('best imaginable caregiving situation'). Higher utility scores thus reflect better care-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Chad Bousman, MPH, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized, individual participant PGx-STaR data will be shared using a controlled-access model. Under this model, the data will be released to a researcher if access criteria are met.
  All requests for data sharing should be made to the Co-Principal Investigators who will be responsible for reviewing and granting requests. Requestors should provide a research proposal for review. In the event that a data sharing request is declined, reasons will be provided to the requestor. If the data sharing request is granted, a data-sharing agreement will be initiated by the Co-Principal Investigators alongside the University of Calgary (lead institution). This agreement will include information on the individual data to be shared; if other documents will be available (e.g., statistical codes, data dictionary), when the data will be available and for how long, and how data access will be provided (e.g., file transfer).
Access Criteria: 1. The requestor is affiliated with an academic institution as an independent investigator or trainee of an independent investigator;
  2. The proposed research question(s) and hypothesis(es) are specific, measurable, and achievable;
  3. The proposed research project will be governed/overseen by a local legal/regulatory body;
  4. The proposed research project poses no risk of invasion of privacy or breaches of confidentiality for trial participants;
  5. A member of the proposed research team has sufficient statistical skills to carry out the proposed analytic plan;
  6. The requestor has sufficient financial and/or human resources to see the proposed research project to completion;
  7. The proposed research question(s) and hypothesis(es) do not conflict with active or planned studies of the Co-Principal Investigators.